CLINICAL TRIAL: NCT02022956
Title: An Open-label, Single-dose Study to Assess the Safety, Tolerability and Pharmacokinetic Properties of BELVIQ in Obese Adolescent Subjects Ages 12-17 (Inclusive)
Brief Title: Single Dose Study to Determine the Safety, Tolerability, and Pharmacokinetic Properties of Lorcaserin Hydrochloride (BELVIQ) in Obese Adolescents From 12 to 17 Years of Age
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APD356-025
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2014-03

CONDITIONS: Pharmacokinetics in Obese Adolescents
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-Label Lorcaserin (BELVIQ) (Experimental)
  Interventions: Drug: Lorcaserin

INTERVENTIONS:
Drug: Lorcaserin
  Other Names: BELVIQ

SUMMARY:
The purpose of this study is to evaluate the PK properties, tolerability, and safety of lorcaserin HCL (BELVIQ) in obese adolescent subjects between the ages of 12 to 17 years old

DETAILED DESCRIPTION:
The purpose is to:

1. Assess the single-dose pharmacokinetic (PK) parameters of lorcaserin and a primary metabolites (M1 and M5) in obese adolescent subjects ages 12-17 (inclusive)
2. Assess the safety and tolerability of a single oral dose of lorcaserin in obese adolescent subjects ages 12-17 (inclusive)

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent subjects aged 12 to 17 years, inclusive at screening
2. a. Eligible female subjects who are sexually active will be:

   * non-pregnant
   * non-lactating
   * agree to continue to use an accepted method of birth control for at least 1 month after study medication administration
3. BMI ≥ 95th percentile for age and gender, but ≤ 44 kg/m21
4. Considered to be in stable health in the opinion of the Investigator.
5. Parent or guardian who can sign written informed consent and subject willing to sign assent

Exclusion Criteria:

1. Clinically significant new illness in the 1 month before screening and any time prior to randomization
2. Significant renal or hepatic disease
3. Secondary (chromosomal, endocrine, or metabolic) causes of obesity
4. Use of medications other than hormonal contraceptives and acetaminophen
5. Use of drugs with serotonergic activity within 1 month before screening
6. Recent treatment with over-the-counter weight loss products or appetite suppressants, or within 3 months of screening and any time prior to randomization with a prescription weight loss drug or lipid dissolving injections or ongoing psychotherapy for weight loss outside of this trial
7. Recent history of alcohol, tobacco, or recreational drug/solvent use
8. Any history of major depression, anxiety, bipolar disorder, schizophrenia, or Axis II psychiatric disease requiring treatment with prescription medication within six months prior to screening

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Assess the single-dose pharmacokinetic (PK) parameters of lorcaserin and a primary metabolites (M1 and M5) in obese adolescent subjects ages 12-17 (inclusive) | 45 min pre-dose and at 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, and 96 hours post-dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Worlwide Clinical Trials, San Antonio, Texas